CLINICAL TRIAL: NCT06444451
Title: A Phase 2, Randomized, Double-blind, Placebo--controlled, Parallel Group, 3-arm, Multinational, Multicenter, Proof-of-concept Study to Evaluate the Efficacy and Safety of Amlitelimab Monotherapy by Subcutaneous Injection in Adult Participants With Severe Alopecia Areata
Brief Title: A Study to Evaluate the Efficacy and Safety of Subcutaneous Amlitelimab Monotherapy Compared With Placebo in Adult Participants With Severe Alopecia Areata
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI18180; 2024-511225-64 (Registry Identifier: CTIS); U1111-1295-6359 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-05-31; First posted 2024-06-05 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Amlitelimab dose group 1 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab
- Amlitelimab dose group 2 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab
- Placebo (Placebo Comparator): Subcutaneous injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlitelimab — Pharmaceutical form: Injection solution Route of administration: SC injection
  Other Names: SAR445229
  Arms: Amlitelimab dose group 1; Amlitelimab dose group 2
Drug: Placebo — Pharmaceutical form: Injection solution Route of administration: SC injection
  Arms: Placebo

SUMMARY:
This is a parallel, Phase 2 multinational, multicenter, randomized, double-blind, placebo-controlled, 3-arm study to investigate the efficacy and safety of subcutaneous (SC) injections of amlitelimab treatment as monotherapy in participants aged 18 years and older with severe alopecia areata (AA). At the end of the double-blind treatment period, all participants will have the option to enter the open-label extension (OLE) period.

The study duration will be up to 160 weeks for participants entering the OLE period including a 2-to-4-week screening, a 36-week randomized double-blind period, an optional OLE period (104 weeks) and a 16-week safety follow-up. The open-label extension period is optional and open to all participants who have completed the double-blind treatment period.

The total number of visits will be up to 38 visits (or 12 visits for those not entering the OLE study).

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of AA of more than 6 months.
* Diagnosis of severe AA, as determined by all of the following:

  1. Hair loss affecting ≥50% of the scalp, as measured by Severity of Alopecia Tool (SALT) at both screening and baseline visits.
  2. Current episode of severe hair loss of less than 8 years. Participants with a history of AA of more than 8 years who have observed episodes of terminal hair regrowth over their scalp ("moving patches" spontaneously or following treatment) in the past 8 years can be included.
  3. Stable disease: no evidence of terminal hair regrowth within 6 months (less than 10% improvement over the past 6 months). (guidance: if participant reports to have quite a bit more hair than 6 months prior, then patient cannot be included).
* Willingness in maintaining a consistent hair style and hair care, including hair products, and to refrain from weaves, extensions, adhesive wigs, other than banded perimeter devices, refrain from shaving of scalp hair for 2 weeks prior to each study visit from baseline to the end of study.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Participants that are currently experiencing other forms of alopecia, including but not limited to: androgenetic alopecia, trichotillomania, telogen effluvium, traction alopecia, scarring alopecia.
* Participants currently with any local or systemic active medical conditions, which in the opinion of the Investigator would interfere with evaluations of the IMP effect on AA due to scalp inflammation, including but not limited to seborrheic dermatitis requiring topical treatment to the scalp, lupus erythematosus, lichen planus, psoriasis, secondary syphilis, tinea capitis, thyroiditis, systemic sclerosis, hair transplants, micropigmentation/tattoo of the scalp.
* Received the specified treatment regimens within the timeframe outlined in the protocol.
* Prior use of any oral JAKi or the topical JAKi ruxolitinib for more than 24 months, regardless if washout period is respected.
* Participants with shaved heads must not enter the study until hair has grown back and SALT score can be reliably administered.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2028-01-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Severity of Alopecia Tool (SALT) score at Week 36 | Baseline to Week 36
  SALT is a quantitative Investigator assessment of AA severity scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss).

SECONDARY OUTCOMES:
Change from the baseline in SALT score at Week 24 (key secondary) | Baseline to Week 24
  SALT is a quantitative Investigator assessment of AA severity scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss).
Proportion of participants achieving a SALT score ≤20 at Weeks 24 and 36 | Week 24 and 36
  SALT is a quantitative Investigator assessment of AA severity scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss).
Time to SALT score ≤20 | Up to Week 36
  SALT is a quantitative Investigator assessment of AA severity scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss).
Proportion of participants achieving a SALT score ≤10 at Weeks 24 and 36 | Week 24 and 36
  SALT is a quantitative Investigator assessment of AA severity scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss).
Time to SALT score ≤10 | Up to Week 36
  SALT is a quantitative Investigator assessment of AA severity scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss).
Proportion of participants achieving a SALT50 at Weeks 24 and 36 | Week 24 and 36
  SALT is a quantitative Investigator assessment of AA severity scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss). SALT50 is 50% reduction from baseline in SALT score.
Proportion of participants achieving a SALT75 at Weeks 24 and 36 | Week 24 and36
  SALT is a quantitative Investigator assessment of AA severity scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss). SALT75 is 75% reduction from baseline in SALT score.
Proportion of participants achieving a SALT90 at Weeks 24 and 36 | Week 24 and 36
  SALT is a quantitative Investigator assessment of AA severity scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss). SALT90 is 90% reduction from baseline in SALT score.
Proportion of participants achieving ClinRO Measure for eyebrow (EB) Hair Loss 0 or 1 with ≥2-point improvement from baseline at Weeks 24 and 36 (among participants with ClinRO Measure for EB Hair Loss ≥2 at Baseline) | Week 24 and 36
  ClinRO Measure for EB Hair Loss is a single item, clinician-reported numeric rating scale (NRS) measuring eyebrow hair loss. Scores range from 0 = normal appearance/no eyebrow hair loss to 3 = severe appearance/severe eyebrow hair loss
Proportion of participants achieving ClinRO Measure for Eyelash (EL) Hair Loss 0 or 1 with ≥2-point improvement from baseline (among participants with ClinRO Measure for EL Hair Loss ≥2 at Baseline) | Week 24 and 36
  ClinRO Measure for EL Hair Loss is a single item, clinician-reported numeric rating scale (NRS) measuring eyelash hair loss. Scores range from 0 = normal appearance/no eyelash hair loss to 3 = severe appearance/severe eyelash hair loss.
Proportion of participants achieving a PGI-C response defined as a score of "moderately improved" or "greatly improved" at Weeks 24 and 36 | Week 24 and 36
  The Patient Global Impression of Change (PGI-C) is a questionnaire that asks participants to provide the overall self-assessment of change in their AA overall on a 5-point scale. The PGI-C will be scored from 1 = Much better to 5 = Much worse.
Proportion of participants achieving a PGI-S response defined as a score of "mild" or "none" at Weeks 24 and 36 | Week 24 and 36
  The Patient Global Impression of Severity (PGI-S) is a single item 5-point scale (1 = no symptoms to 5 = very severe symptoms) which asks a participant to assess current severity of AA symptoms.
Mean changes from baseline in SKINDEX-16AA at Weeks 24 and 36 | Baseline to Week 24 and 36
  Skindex-16 for alopecia areata (SKINDEX-16AA) is a tool used to assess the health-related quality of life in participants with skin disorders. The score ranges from 0 to 100, with higher scores indicating a greater burden of AA on the patient.
Proportion of participants with PRO Scalp Hair Assessment score of 0 to 1 with ≥2-point improvement from baseline (among participants with PRO Scalp Hair Assessment score ≥3 at Baseline) | Week 24 and 36
  Scalp Hair Assessment patient reported outcome (PRO) is a single item, patient-reported NRS using a 5-point response scale and ranging from 0 to 4, with 0 = no missing hair (0% scalp hair missing) and 4 = nearly all or all missing hair (95- 100% scalp hair missing).
Proportion of participants achieving grade 0 or 1 with ≥2-point improvement from baseline PRO Measure for EB Hair Loss (among participants with PRO Measure for EB Hair Loss ≥2 at Baseline) | Week 24 and 36
  PRO Measure for Eyebrow Hair Loss™ is a single item, patient-reported NRS measuring eyebrow hair loss, ranging from 0 to 3, with 0 = full coverage/no eyebrow hair loss and 3 = barely any/no notable eyebrow hair.
Proportion of participants achieving grade 0 or 1 with ≥2-point improvement from baseline PRO Measure for EL Hair Loss at Weeks 24 and 36 (among participants with PRO Measure for EL Hair Loss ≥2 at Baseline) | Week 24 and 36
  PRO Measure foe Eyelash Hair Loss™ is a single item, patient-reported NRS measuring eyelash hair loss, ranging from 0 to 3, with 0 = full coverage/no eyelash hair loss and 3 = barely any/no notable eyelash hair.
Proportion of participants who experienced treatment-emergent adverse events (TEAEs), experienced treatment-emergent serious adverse event (TESAEs) and/or Treatment-Emergent adverse event of special interest (AESIs) | Up to week 156
Serum amlitelimab concentrations measured at prespecified timepoints | Up to Week 156
Incidence of ADAs of amlitelimab at prespecified timepoints | Up to Week 156

CONTACTS AND LOCATIONS:
Locations (74):
- United States (17):
  - Total Skin and Beauty Dermatology Center- Site Number : 8400018, Birmingham, Alabama
  - First OC Dermatology- Site Number : 8400014, Fountain Valley, California
  - Center for Dermatology Clinical Research- Site Number : 8400008, Fremont, California
  - UC Irvine Healthcare - Gottschalk Medical Plaza- Site Number : 8400007, Irvine, California
  - Dermatology Research Associates - Los Angeles- Site Number : 8400015, Los Angeles, California
  - New Horizon Research Center- Site Number : 8400017, Miami, Florida
  - Dawes Fretzin Clinical Research- Site Number : 8400010, Indianapolis, Indiana
  - Michigan Center for Research Company- Site Number : 8400016, Clarkston, Michigan
  - Joel Schlessinger, PC- Site Number : 8400021, Omaha, Nebraska
  - Icahn School of Medicine at Mount Sinai- Site Number : 8400003, New York, New York
  - DJL Clinical Research - Charlotte - Park Road- Site Number : 8400013, Charlotte, North Carolina
  - Cleveland Clinic- Site Number : 8400028, Cleveland, Ohio
  - Apex Clinical Research Center- Site Number : 8400027, Mayfield Heights, Ohio
  - Vital Prospects Clinical Research Institute - Tulsa- Site Number : 8400004, Tulsa, Oklahoma
  - Oregon Medical Research Center- Site Number : 8400002, Portland, Oregon
  - Health Concepts- Site Number : 8400001, Rapid City, South Dakota
  - Progressive Clinical Research - San Antonio- Site Number : 8400019, San Antonio, Texas
- Argentina (3):
  - Investigational Site Number : 0320002, Rosario, Santa Fe Province
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
- Australia (2):
  - Investigational Site Number : 0360001, Sydney, New South Wales
  - Investigational Site Number : 0360003, Melbourne, Victoria
- Investigational Site Number : 1000001, Sofia, Bulgaria
- Canada (5):
  - Investigational Site Number : 1240005, Calgary, Alberta
  - Investigational Site Number : 1240007, Calgary, Alberta
  - Investigational Site Number : 1240001, Winnipeg, Manitoba
  - Investigational Site Number : 1240003, Hamilton, Ontario
  - Investigational Site Number : 1240006, Markham, Ontario
- Chile (4):
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
- China (3):
  - Investigational Site Number : 1560022, Chengdu
  - Investigational Site Number : 1560006, Hangzhou
  - Investigational Site Number : 1560001, Shanghai
- Czechia (3):
  - Investigational Site Number : 2032104, Ostrava
  - Investigational Site Number : 2030011, Prague
  - Investigational Site Number : 2030012, Prague
- France (4):
  - Investigational Site Number : 2500001, Brest
  - Investigational Site Number : 2500002, Nice
  - Investigational Site Number : 2500003, Paris
  - Investigational Site Number : 2500004, Rouen
- Germany (6):
  - Investigational Site Number : 2760006, Augsburg
  - Investigational Site Number : 2760008, Berlin
  - Investigational Site Number : 2760007, Berlin
  - Investigational Site Number : 2760001, Hamburg
  - Investigational Site Number : 2760003, Münster
  - Investigational Site Number : 2760004, Osnabrück
- Italy (4):
  - Investigational Site Number : 3800004, Milan, Milano
  - Investigational Site Number : 3800003, Naples, Napoli
  - Investigational Site Number : 3800002, Rome, Roma
  - Investigational Site Number : 3800001, Bologna
- Japan (7):
  - Investigational Site Number : 3920003, Ebina-shi, Kanagawa
  - Investigational Site Number : 3920001, Yokohama, Kanagawa
  - Investigational Site Number : 3920002, Kamiamakusa, Kumamoto
  - Investigational Site Number : 3920005, Koto-ku, Tokyo
  - Investigational Site Number : 3920004, Fukuoka
  - Investigational Site Number : 3920006, Tokyo
  - Investigational Site Number : 3920001, Yokohama
- Investigational Site Number : 5280004, Rotterdam, Netherlands
- Investigational Site Number : 6420001, Cluj-Napoca, Romania
- Spain (7):
  - Investigational Site Number : 7240005, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240010, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240007, Pozuelo de Alarcón, Madrid
  - Investigational Site Number : 7240004, Alicante
  - Investigational Site Number : 7240002, Córdoba
  - Investigational Site Number : 7240006, Madrid
  - Investigational Site Number : 7240008, Madrid
- United Kingdom (6):
  - Investigational Site Number : 8260003, London, London, City of
  - Investigational Site Number : 8260004, Salford, Manchester
  - Investigational Site Number : 8260006, Oxford, Oxfordshire
  - Investigational Site Number : 8260005, Dundee
  - Investigational Site Number : 8260007, London
  - Investigational Site Number : 8260001, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DRI18180 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25760&tenant=MT_SNY_9011